CLINICAL TRIAL: NCT05517902
Title: A Phase 3 Multicenter, Single-Arm, Open-Label Study Evaluating the Safety, Tolerability and Efficacy of StrataGraft® Construct in Pediatric Subjects With Deep Partial Thickness (DPT) Thermal Burns
Brief Title: StrataGraft Safety, Tolerability and Efficacy in Pediatric Subjects
Acronym: StrataSTEPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNK15011001
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Skin Wound; Burns; Trauma-related Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2 to < 12 years Age Group Cohort (Experimental): Single application of StrataGraft to 0.5% to 10% total body surface area (TBSA) on Day 1.
  Interventions: Biological: StrataGraft
- 12 to ≤ 17 years Age Group Cohort (Experimental): Single application of StrataGraft to 0.5% to 10% TBSA on Day 1.
  Interventions: Biological: StrataGraft

INTERVENTIONS:
Biological: StrataGraft — StrataGraft® Construct

SUMMARY:
Autografting is a surgical procedure to transplant healthy skin (donor skin) from another part of the participant's own body (donor site) to the burned part. Autografting is the usual treatment for DPT burns.

It works to close the wound, but can cause other problems:

* Donor sites are painful, can become infected or scarred, or can even become full thickness (FT) wounds themselves
* Treatment problems can require more grafting
* Additional surgery increases the risk of medical problems caused by the treatment

Stratatech is trying to find a safe and effective alternative to autografting to promote the healing of severe burns. The purpose of this study was to evaluate whether StrataGraft treatment eliminates or reduces the need for autografting and promotes wound closure in a pediatric population with thermal burns that contain intact dermal elements and for which autografting is clinically indicated (DPT burns).

Participants were enrolled into one of two age-based cohorts: 2 to < 12 years and 12 to ≤ 17 years to receive a single application of StrataGraft, in up to 3 non-contiguous DPT burn areas located on the same extremity or plane of the torso.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the parent(s) or legal guardian(s) and assent from the child when appropriate
* Have enough healthy skin to reserve as donor site(s), in case autografting becomes necessary
* Thermal burns of no more than a total of 30% TBSA
* Study treatment sites that are DPT in depth and which are clinically indicated for excision and autografting, and located on the torso or extremities
* Study treatment area(s) totaling 0.5% to 10% TBSA and may be composed of up to 3 non-contiguous areas located on the same extremity or plane of the torso
* Sufficient healthy skin available and reserved as a donor site in the event that the StrataGraft treatment site requires autografting

Exclusion Criteria:

* Is pregnant or breastfeeding
* Receiving treatment to suppress the immune system and/or systemic corticosteroids (inhaled corticosteroids are permitted)
* A known history of malignancy
* Pre-admission insulin-dependent diabetes
* Concurrent trauma, conditions, and/or personal situations that, in the opinion of the investigator, may compromise the participant's safety or the study objectives
* A burn injury that occurred ≥ 14 days prior to planned StrataGraft application Is expected to survive less than 12 months
* Is participating in another interventional trial, or did within 90 days before enrollment
* A proposed study treatment site that has been previously excised or autografted; located adjacent to an undebrided/unexcised burn area; demonstrates signs and symptoms of wound infection, per judgement of the clinical investigator; lies across joints or is located on the feet (i.e., distal to the malleolus), hands (distal to the wrist), face, neck, buttocks, perineum, or genitalia

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Stratatech, a Mallinckrodt Company
Locations (1):
- Research Site, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant took part in the study at a single clinical site in the United States from 28 April 2023 to 9 May 2024.
Period: Overall Study
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled and received StrataGraft.
Groups:
- 2 to < 12 Years Age Group Cohort; 12 to ≤ 17 Years Age Group Cohort: Single application of StrataGraft to 0.5% to 10% TBSA on Day 1.
- Total: Total of all reporting groups
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Confirmed Complete Closure of StrataGraft Treatment Sites Without Autograft Within 12 Weeks of StrataGraft Application
Description: Confirmed complete wound closure is defined as complete skin re-epithelialization confirmed at 2 consecutive visits at least 2 weeks apart, but no later than Week 20. Percentage of participants whose burn healed after StrataGraft treatment without needing the doctor to treat the burn with skin cut from other parts of the patient's own body were reported.
Time Frame: Up to Week 12
Population: Safety population included all participants who were enrolled and received StrataGraft.
Measure: Number; unit: percentage of participants
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort
Number analyzed (Participants) | 1 | 0
percentage of participants | 100 |

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant who is administered a study treatment, which does not necessarily have to have a causal relationship with this treatment. TEAEs are AEs with an onset date on or after the start of StrataGraft treatment.
Time Frame: Up to Month 12
Population: Safety population included all participants who were enrolled and received StrataGraft.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort
Number analyzed (Participants) | 1 | 0
Participants | 1 |

3. Secondary Outcome: Percentage of StrataGraft Treatment Sites Per Participant Closed at Week 12 Without Autograft Placement
Description: Wound closure was evaluated through visual inspection by the investigator. Complete wound closure was defined as "complete re-epithelialization of the wound without drainage," confirmed at 2 consecutive visits at least 2 weeks apart.
Time Frame: At Week 12
Population: Safety population included all participants who were enrolled and received StrataGraft.
Measure: Number; unit: percentage of treatment sites
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort
Number analyzed (Participants) | 1 | 0
percentage of treatment sites | 100 |

4. Secondary Outcome: Number of Confirmed Complete Wound Closures of the StrataGraft Treatment Sites on or Before Week 12 Without Autograft Placement
Description: Complete wound closure was defined as "complete re-epithelialization of the wound without drainage," confirmed at two consecutive visits at least two weeks apart.
Time Frame: Up to Week 12
Population: Safety population included all participants who were enrolled and received StrataGraft.
Measure: Number; unit: number of complete wound closure
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort
Number analyzed (Participants) | 1 | 0
number of complete wound closure | 1 |

5. Secondary Outcome: Mean of Averaged Percent Area of StrataGraft Treatment Sites Per Participant Autografted by Week 12
Time Frame: Up to Week 12
Population: Safety population included all participants who were enrolled and received StrataGraft. None of the participant had StrataGraft treatment site that required autografting.
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Safety population included all participants who were enrolled and received StrataGraft.
Arm/Group | 2 to < 12 Years Age Group Cohort | 12 to ≤ 17 Years Age Group Cohort
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 to < 12 Years Age Group Cohort (N=1) | 12 to ≤ 17 Years Age Group Cohort (N=0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
This study had low accrual and only 1 participant was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT05517902/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan_Memo (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT05517902/SAP_001.pdf